CLINICAL TRIAL: NCT06216132
Title: A Phase 1, Placebo-controlled, Single-Ascending-Dose, Study of BIOPIN 6 in Healthy Adults
Brief Title: Study of the BIOPIN 6 Naltrexone Implant in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akyso Therapeutics, LLC (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Laboratory Corporation of America (Industry); Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIOPIN101; 5UG3DA048338-02 (NIH)
Record Dates: First submitted 2023-12-27; First posted 2024-01-22 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: Determine naltrexone and 6b-naltrexole pharmacokinetic parameters in subjects administered a single dose of BIOPIN 6 [BIOPIN 6 implants containing 4.8g (dose-level #1) or 9.6g (dose-level #2) naltrexone]. Each of the two dose groups will be compared to a placebo implant group. The initial study design had 3 groups and a high dose group receiving 14.4 g naltrexone. After the PK data became available for the second cohort, the sponsor chose to not proceed with the final cohort because the target PK parameters had been achieved with the 9.6 gram group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The surgeon and the team performing the subcutaneous implant and removal will be unmasked. All other staff and subjects will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BIOPIN-6 active implant (Experimental): Two sequential cohorts receiving 4.8 or 9.6 BIOPIN 6 implanted into a subcutaneous pocket in the upper abdominal wall.
  Interventions: Combination Product: BIOPIN-6 Active Implant with Naltrexone
- BIOPIN-6 placebo implant (Placebo Comparator): The placebo will be an implant consisting of the poly-d-l Lactic Acid and polycaprolactone contained in BIOPIN 6 without naltrexone.
  Interventions: Device: BIOPIN-6 Placebo Implant

INTERVENTIONS:
Combination Product: BIOPIN-6 Active Implant with Naltrexone — An extended release formulation of naltrexone implanted in the subcutaneous space.
  Other Names: BIOPIN; Subcutaneous naltrexone implant; Extended release naltrexone implant
  Arms: BIOPIN-6 active implant
Device: BIOPIN-6 Placebo Implant — The placebo will be an implant consisting of the poly-d-l Lactic Acid and polycaprolactone contained in BIOPIN 6 without naltrexone.
  Arms: BIOPIN-6 placebo implant

SUMMARY:
The purpose of this study is to evaluate the safety and blood levels of a medicine, naltrexone, contained within an implant in healthy volunteers age 18 to 65 years. To do this, the implant containing the drug will be inserted under the skin, left in place for 3 months and then removed.

DETAILED DESCRIPTION:
Naltrexone (NTX) is a medication that helps people with opioid and alcohol dependence. It works by blocking the effects of opioids like heroin in the body. In the United States, participants can get NTX in two forms: a pill participants take once a day (Revia) and a shot participants get once a month (Vivitrol). Even though NTX is good at stopping the effects of opioids, some people find it hard to take it regularly. That's why scientists are looking into making a new version of NTX that participants only need to take once a month. This could make it easier for people with opioid use problems to stick with their treatment plan.

The device being tried out in this research is called BIOPIN-6. It's made to stay in the body for more than a month. The study will go on for three months and aims to check if the BIOPIN-6 is safe and how much medicine it releases into the blood. Once the three months are up, the device will be taken out.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included in the study:

* Healthy male or female volunteer, aged 18-to-55 years, inclusive.
* BMI must be between 18 and 32 kg/m2 (inclusive) and weigh a minimum of 50 kg (110 lbs).
* If female, be postmenopausal (at least 2 years prior to dosing) or agree to use an acceptable form of birth control from screening until 12 weeks after dosing. Subjects who claim postmenopausal status will have status confirmed with a follicle stimulating hormone (FSH) test. Acceptable forms of birth control for females include the following:

  * Vasectomized partner (at least 6 months prior to dosing)
  * Surgical sterilization (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) at least 6 months prior to dosing
  * Non-surgical permanent sterilization (eg, Essure procedure) at least 3 months prior to dosing.
  * Abstinence (must agree to use a double barrier method if they become sexually active during the study)
  * Double barrier (diaphragm with spermicide; condoms with spermicide)
  * Oral hormonal contraceptives
* Not Breast feeding
* Negative tests for human immunodeficiency virus (HIV), Hepatitis C antibody, Hepatitis B surface antigen, and Covid
* Able and willing to comply with the requirements of the protocol
* Able and willing to provide written informed consent
* Willing to undergo a minor surgical procedure under local anesthetic to allow for investigational drug administration in the subcutaneous tissue
* Agree to avoid blunt trauma to the implantation site
* Agree that after implantation, not to shower for 2 days and not to bathe/swim for 4 weeks

Exclusion Criteria:

Subjects must have none of the exclusion criteria to be included in the study.

* Clinically significant abnormal finding on the physical exam, medical history, electrocardiogram (EKG), or clinical laboratory results at screening. In particular, values of liver function tests (ALT, AST, bilirubin, albumin, GGT) and kidney function tests (creatinine, blood urea nitrogen) and reticulocytes shall not deviate by more than 25% from the ranges of normal.
* Blood pressure: systolic >140 mmHg, diastolic >90 mmHg. [Europe Soc Hypertension guidelines]
* Heart rate: >100 beats/minute.
* Hemoglobin for female <11.5 and for male <12.5 are excluded.
* Have a known or suspected history or family history of adverse reactions or hypersensitivity to the study drugs or to drugs with a similar chemical structure.
* History or presence of gastrointestinal, hepatic or renal disease, or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Is on anticoagulant medications other than aspirin or NSAIDs. Agree to stop aspirin or NSAIDs 1 week prior to Biopin 6 implantation
* Used any over-the-counter (OTC) medication, nutritional or dietary supplements, herbal preparations, or vitamins within 7 days prior to the first dose of medication.
* Used any prescription medication within 14 days prior to the first dose of study medication.
* More than moderate drinking averaged over the last month as assessed by history:

  o Moderate drinking is here defined as up to 3 drinks per week. The standard drink will be defined by the guidelines of the National Institute on Alcohol Abuse and Alcoholism (NIAAA) and will contain no more than 14 g of alcohol.
* Smoking: Use of tobacco or nicotine-containing products within the 3-month period preceding study drug administration is exclusionary.
* Positive urine drug screen for amphetamines, barbiturates, benzodiazepines, cocaine, opiates, cannabinoids, phencyclidine, propoxyphene, methadone, methaqualone, and alcohol at the screening and Day -1 tests.
* Any methadone use 14 days prior to screening, and up to Study Day -1.
* Has had a naltrexone implant in the past 24 months.
* Has received treatment with an extended naltrexone product (e.g. Vivitrol) in the past 12 months.
* Fails the naloxone challenge test
* Has a condition which requires treatment with opioid based medication.
* Has a known hypersensitivity to naltrexone.
* Has a known hypersensitivity to materials based on poly-d-l Lactic Acid and polycaprolactone (e.g. biodegradable sutures, surgical implants or previous biodegradable implants).
* Has a known hypersensitivity to local anesthesia.
* Is prone to skin rashes, irritation or has a skin condition such as recurrent eczema that is likely to impact the implant site area, or as determined by the evaluating physician.
* Is known to form keloids at the site of skin injury.
* Demonstrates any abnormal skin tissue in the proposed implantation area
* Previous surgery to the upper abdominal wall
* Donated blood or plasma within 30 days prior to the first dose of study medication.
* Participated in another clinical trial within 30 days prior to the first dose of study medication.
* Is participating or intending to participate in any other clinical trial during the duration of this study.
* Any elevated risk for suicide measured using the Columbia Suicide Severity Rating Scale, endorsing any of the items in the past month (C-SSRS, Lifetime)
* Not as much as "mild" depression as measured by the HAM-D17 test: HAM-D17 score must be 0-10.
* Any additional condition(s) that in the investigator's opinion would prohibit the participant from completing the study or would not be in the best interest of the participant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Naltrexone plasma levels (average) | Day 0 to Day 98
  Naltrexone Area under the plasma concentration versus time curve (AUC) [(ng/ml) x hr]
Naltrexone plasma levels (peak) | Day 0 to Day 98
  Naltrexone Peak Plasma Concentration (Cmax) [ng/ml]
Naltrexone plasma levels (peak onset) | Day 0 to Day 98
  Naltrexone time to peak plasma concentration (Tmax) [hr]
6-b-natlrexol plasma levels | Day 0 to Day 98
  6-b-naltrexol Area under the plasma concentration versus time curve (AUC) [(ng/ml) x hr]
6-b-natlrexol plasma levels (peak) | Day 0 to Day 98
  6-b-naltrexol Peak Plasma Concentration (Cmax) [ng/ml]
6-b-natlrexol plasma levels (time to onset of peak)) | Day 0 to Day 98
  6-b-naltrexol time to peak plasma concentration (Tmax) [hr]

SECONDARY OUTCOMES:
Adverse events | Day 0 to Day 98
  Number of participants with adverse events as assessed by CTCAE v5.
Clinical laboratory values | Day 0 to Day 98
  Number of participants with laboratory abnormalities as assessed by CTCAE v5.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bertoch, MD, Principal Investigator — Cenexel JBR
Locations (1):
- JBR Clinical Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No